CLINICAL TRIAL: NCT01541007
Title: A Randomized, Open Label, Multicenter, Phase II Trial Comparing The Conventional 3 Weekly Schedule Of Cabazitaxel With A Weekly Regimen In Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: A Study Looking at Novel Scheduling of Cabazitaxel for Patients With Metastatic Prostate Cancer
Acronym: ConCab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey Yachnin M.D., PhD. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Yachnin M.D., PhD., Director Clinical Trials Unit, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-004178-27
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Prostate Cancer; Metastatic; Castration Resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Cabazitaxel Schedule (Active Comparator): Cabazitaxel 25 mg/m2 every three weeks
  Interventions: Drug: Cabazitaxel
- Weekly cabazitaxel schedule (Experimental): cabazitaxel 10 mg/m2 given weekly for 5 consecutive weeks of a six week cycle
  Interventions: Drug: weekly cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 25 mg/m2 every three weeks
  Arms: Standard Cabazitaxel Schedule
Drug: weekly cabazitaxel — 10 mg/m2 dag 1,8,15,22. Cycle length is 6 weeks
  Arms: Weekly cabazitaxel schedule

SUMMARY:
Cabazitaxel has shown significant efficacy as second line chemotherapy after Docetaxel in men with metastatic castration resistant prostate cancer. This was demonstrated in the Tropic Study where Cabazitaxel showed survival superiority compared to mitoxantrone. Almost one in 4 patients treated with Cabazitaxel in this study required dose reductions or dose delays or stopped treatment due to toxicity. ConCab examines another scheduling for cabazitaxel to see if we can improve tolerability so that patients will receive a higher percentage of the treatment as planned.

DETAILED DESCRIPTION:
ConCab compares the standard treatment of cabazitaxel 25 mg/m2 every three weeks with an experimental scheduling of 10 mg/m2 for 5 consecutive weeks of a 6 week cycle. In both study arms the planned cumulative dose of cabazitaxel at week 18 is 150 mg/m2. Our study aims to evaluate differences in the total received dose in relation to the planned dose as a measure of which of the 2 treatment schedules is superior.

ELIGIBILITY:
Inclusion Criteria:¨

* Histological confirmed prostate cancer
* Macroscopic metastatic disease
* Prior treatment with Docetaxel
* Castration resistant disease defined as:Serum testosterone (< 0.5 ng/ml) and:
* Increase in measurable disease (RECIST 1.1, see appendix 10) or
* For non-measurable disease, the appearance of at least one new lesion on nuclear scintigraphy) or
* A rising PSA from the previous reference value on 2 consecutive occasions at least one week apart
* Written informed consent

Exclusion Criteria:

* Less than 21 days since prior treatment with chemotherapy
* Less than 14 days since radiotherapy or surgery to the start of cabazitaxel - Less than 4 weeks after stopping endocrine therapies including antiandrogen, abiraterone or other new agents.
* Prior isotope therapy or radiotherapy to > 30% of bone marrow (whole pelvic radiotherapy is not an exclusion criteria)
* Persistent adverse events from previous cancer therapies > grade 1 (CTCAE - Version 4.0) with the exception of alopecia. (With respect to peripheral neuropathy and nail changes grade 2 is acceptable)
* ECOG performance status > 1
* Known CNS malignancy
* Within 6 months of randomization:

  * myocardial infarction,
  * unstable angina,
  * angioplasty,
  * bypass surgery,
  * stroke,
  * TIA, or
  * congestive heart failure NYHA class III or IV
* Within 3 months prior to randomization:

  * treatment resistant peptic ulcer disease,
  * infectious or inflammatory bowel disease,
  * pulmonary embolism
  * Any severe acute or chronic medical condition that places the patient at increased risk of serious toxicity or interferes with the interpretation of study results
* History of hypersensitivity to docetaxel or polysorbate 80
* Inadequate organ and bone marrow function as evidenced by:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count < 1.5 x 109/L,
  * Platelet count < 100 x 109/L,
  * AST/SGOT and/or ALT/SGPT > 1.5 x ULN;
  * Total bilirubin > 1.0 x ULN,
  * Serum creatinine > 1.5 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance < 60 mL/min should be excluded (http://mdrd.com/ for on-line calculation)
* Concurrent or planned treatment with potent inhibitors or inducers of cytochrome P450 3A4/5. A one week wash out period is necessary for patients who are already on these treatments.
* Patients with reproductive potential not implementing accepted and effective method of contraception.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Relative cumulative dose of cabazitaxel at week 18 | week 18 after start of treatment
  The primary endpoint compares the cumulative dose of cabazitaxel that is received relative to the planned dose at 18 weeks of therapy. The cumulative dose of cabazitaxel in relation to the expected dose is a reflection of both tolerability and efficacy. Patients stopping treatment due to disease progression prior to week 18 will have lower relative cumulative doses as will patients with poor tolerability due to dose reductions and delays.

SECONDARY OUTCOMES:
Overall Survival | when the last enrolled patient has completed 18 weeks of therapy or has stopped therapy at an earlier date
  Overall survival is defined as the length of time from randomization to death from any cause
Progression free survival | when the last enrolled patient has completed 18 weeks of therapy or has stopped therapy at an earlier date
  Progression free survival is defined as the length of time from randomisation to the first documentation of one of the following: PSA progression or pain progression or death due to any cause or radiological disease progression
PSA Response | when the last enrolled patient has completed 18 weeks of therapy or has stopped therapy at an earlier date
  Only considered after 12 weeks of treatment. PSA response is defined as a 50% or greater decline in serum PSA from baseline given that baseline PSA is at least 10 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Yachnin, MD, PhD, Study Chair — Karolinska University Hosptial
Locations (1):
- Deapartment of Oncology Karolinska University Hospital, Stockholm, Sweden